CLINICAL TRIAL: NCT03331848
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-arm Phase IIa Trial to Evaluate the Efficacy, Safety, and Tolerability of 8-week Oral Treatment With PXT002331 (Foliglurax) in Reducing Levodopa-Induced Dyskinesia and Wearing OFF in Subjects With Parkinson's Disease Experiencing Motor Complications of Levodopa Therapy (ATTUNED)
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of PXT002331 (Foliglurax) in Reducing Levodopa-Induced Dyskinesia and Wearing OFF in Subjects With Parkinson's Disease Experiencing Motor Complications of Levodopa Therapy (ATTUNED)
Acronym: ATTUNED
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Prexton Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PXT-CL17-003
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2017-10

CONDITIONS: Parkinson Disease
Keywords: Levodopa-Induced Dyskinesia (LID); Foliglurax; Parkinson's Disease; mGlu4 PAM
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PLACEBO (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- PXT002331 - 20mg (Experimental)
  Interventions: Drug: PXT002331 - 20mg

INTERVENTIONS:
Drug: Placebo oral capsule — BID
  Arms: PLACEBO
Drug: PXT002331 - 20mg — Oral
  Arms: PXT002331 - 20mg

SUMMARY:
This is a Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-arm Phase IIa proof of concept in subjects with PD treated with a stable dose of levodopa who are experiencing Motor Complications of Levodopa Therapy

ELIGIBILITY:
Inclusion Criteria:

* Between 35 and 85 years of age, inclusive, at the time of signing informed consent
* Diagnosed after the age of 30 years with idiopathic PD
* A documented medical history of idiopathic PD for at least 3 years
* Disease severity of 2 to 4 on the modified Hoehn and Yahr scale when in the OFF state
* Been treated with a stable regimen of levodopa-containing therapy
* Subjects must be receiving at least 3 doses per day of levodopa-containing therapy, and must be on a stable dose for at least 2 weeks for immediate-release levodopa or at least 6 weeks for prolonged-release levodopa preparations prior to the first screening visit
* Experienced LID over a period of at least 3 months prior to randomization
* If needed, in the opinion of the investigator, subjects must have a caregiver
* Female subjects will be women of non-childbearing potential

Exclusion Criteria:

* Patient is currently participating in or has participated in another study in the last 3 months
* Subjects with atypical, secondary, or drug-induced Parkinsonism
* Subjects with a history of dyskinesia that was exclusively diphasic, OFF state, myoclonic, dystonic, or akathetic without peak-dose dyskinesia
* Subjects with a MoCA score of <25
* Subjects who have, or who had a history of, any clinically significant hepatic or gallbladder disorder, as determined by the investigator
* Subjects who have dementia, currently active psychosis, or hallucinations.
* Suicide attempt within 1 year prior to the first screening visit, or severe suicidal ideation within 6 months prior to the first screening visit
* Subject has a current diagnosis of epilepsy,
* Any known contraindication to the use of levodopa, including a history of malignant melanoma or a history of narrow-angle glaucoma
* Carcinoma or successfully treated squamous cell carcinoma of the skin and no sing of disease recurrence for at least 5 years
* Subjects who have had a clinically significant illness within 4 weeks before the first dose, as determined by the investigator
* Subjects with scheduled surgeries/hospitalizations during the study period
* Any advanced, severe, or unstable disease (other than PD) that may interfere with the primary and secondary study outcome evaluations
* Subjects who have undergone prior neurosurgical operation for PD,
* Subjects currently taking (or expected to be administered during the course of the study) any of the prohibited medications (amantadine, safinamide, dopamine-antagonists).

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Unified Dyskinesia Rating Scale (UDysRS) total score in subjects with PD experiencing levodopa-induced dyskinesia. | 26 days